CLINICAL TRIAL: NCT01349426
Title: Standard Stapling Technique Versus Bipolar Fusion (With The Ligasure Impact and Force Triad Generator) To Complete The Fissure During Major Lung Resection: A Prospective Randomized Controlled Trial
Brief Title: Ligasure II: Standard Stapling Versus Ligasure
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: diffculty to include patients
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1008067; 2010-A00666-33 (Other: AFSSAPS registration)
Record Dates: First submitted 2011-05-04; First posted 2011-05-06 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Lung Resection
Keywords: Lung resection; Parenchymal pneumostasis, haemostasis; Fissure closure; Automatic staplers,LigaSure, Force Triad Generator; Bipolar fusion; Procedure cost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LigaSure (Experimental): * Arm 1
  * Patients undergoing lung surgery
  Interventions: Device: LigaSure Force Triad Vessel Sealing System
- Automatic Staplers (Active Comparator): * Arm 2
  * Patients undergoing lung surgery
  Interventions: Device: LigaSure Force Triad Vessel Sealing System

INTERVENTIONS:
Device: LigaSure Force Triad Vessel Sealing System — Quality of parenchymal pneumostasis comparison after fissure closure: LigaSure vs automatic staplers
  Other Names: Automatic Staplers TA30P, TA55; Endo GIA II MULTIFIRE

SUMMARY:
Surgical staplers have become standard for ligation, division, resection, anastomosis and closure in many surgical procedures. Staplers are utilized in thoracic surgery routinely for pulmonary parenchymal resection and closure, ligation of vessels and bronchi. In addition, closure of incomplete fissure/s is a frequent need in pulmonary surgery. Although generally safe and efficacious, staplers and staple loads are expensive, and can result in micro air leaks. The LigaSure Vessel Sealing System presents as a potentially faster and less expensive alternative to staplers. The LigaSure Vessel sealing system utilizes a combination of heat generated via bi-polar radiofrequency energy and precise jaw pressure to denature the collagen and elastin in tissue and blood vessels. The newly released Force Triad Generator and the Impact, a 10 mm jaw sealing device (Ligasure system, COVIDIEN Society) may offer improved performance in terms of tissue sticking due to an improved sealing algorithm, and to the jaw configuration of the Impact. The study main objective is to compare the quality of parenchymal pneumostasis after fissure closure achieved with staplers vs that achieved with LigaSure.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years
* Patients scheduled for thoracotomy, lobectomy or bilobectomy
* Patients must give informed consent

Exclusion Criteria:

* Patient is unwilling or unable to provide informed consent
* Patients who can not tolerate thoracotomy
* Patients who require extensive dissection to release adhesions which may result in air leak and/or bleeding unrelated to the quality of the parenchymal seal achieved by the devices in question
* Patients with no parenchymal bridge between lobes; 100% complete fissure.
* Patients with complete incomplete fissure with a thickness > 1.5 cm measure intraoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2010-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Rates of post-operative air leak between the two techniques | Day 1

SECONDARY OUTCOMES:
Compare the number of lung stitches between LigaSure device and standard staplers | Day 1
Evaluate the cost of LigaSure vs standard staplers in similar procedures including the cost of each instrument and the staple loads fired. | Day 1

CONTACTS AND LOCATIONS:
Overall Officials: TIFFET Olivier, MD, Principal Investigator — CHU Sainte-Etienne
Locations (10):
- France (10):
  - CHU Lyon-Department of Thoracic Surgery, Cardiovascular and Chest Hospital, Bron
  - CHU Clermont Ferrand - Service of Thoracic Surgery, Clermont-Ferrand
  - CHU Grenoble - Department of Vascular and Thoracic Surgery, Grenoble
  - CHU Lille - Service of Thoracic Surgery, Lille
  - Hospital Dupuytren - Department of Thoracic and CardioVascular Surgery, Limoges
  - CHU Marseille - Department of Thoracic Surgery, Marseille
  - CHU Nice - Pasteur Hospital - Department of Thoracic Surgery, Nice
  - Chu Saint-Etienne, Saint-Etienne
  - CHU Strasbourg - Service of Thoracic Surgery, Strasbourg
  - Department of Thoracic Surgery, Hospital Larrey, CHU Toulouse, Toulouse